CLINICAL TRIAL: NCT00077532
Title: A Study of Intra-Patient Escalating Doses of MDX-010 Given Alone or in Combination With Two gp100 Peptides Emulsified With Montanide ISA-51 in the Treatment of Patients With Stage IV Melanoma
Brief Title: Monoclonal Antibody With or Without gp100 Peptides Plus Montanide ISA-51 in Treating Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 040083; 04-C-0083; MDX-010-19; NCI-6532; CDR0000352187; NCT00076167 (obsolete NCT alias)
Record Dates: First submitted 2004-02-10; First posted 2004-02-12 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — incomplete Freund's adjuvant; Ipilimumab

INTERVENTIONS:
Biological: gp100 antigen
Biological: incomplete Freund's adjuvant
Biological: ipilimumab

SUMMARY:
RATIONALE: Biological therapies, such as MDX-010, work in different ways to stimulate the immune system and stop tumor cells from growing. Vaccines made from gp100 peptides may make the body build an immune response to kill tumor cells. Combining the vaccines with Montanide ISA-51 may cause a stronger immune response and kill more tumor cells. It is not yet known whether monoclonal antibody therapy is more effective with or without vaccine therapy in treating advanced melanoma.

PURPOSE: This randomized phase II trial is studying monoclonal antibody therapy alone to see how well it works compared to monoclonal antibody therapy, gp100 peptides, and Montanide ISA-51 in treating patients with stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the clinical response in patients with stage IV melanoma treated with escalating doses of anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody (MDX-010) with or without gp100 peptides emulsified in Montanide ISA-51.

Secondary

* Determine the safety and toxicity profile of these regimens in these patients.
* Determine the immunologic response in patients treated with these regimens.
* Determine the pharmacokinetics of these regimens in these patients.
* Determine, in HLA-A*0201-positive patients, the differences in responses between patients previously vaccinated with gp100 peptides and patients not previously vaccinated.

OUTLINE: This is a 2-part, partially randomized study.

* Part I (closed as of 3/7/2005):

  * HLA-A*0201-negative patients: Patients receive anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody (MDX-010) IV over 90 minutes on day 1. Treatment repeats every 3 weeks for up to 6 doses (3 courses of 3 escalating doses) in the absence of disease progression or unacceptable toxicity.
  * HLA-A*0201-positive patients: Patients are stratified according to prior exogenous gp100 peptide immunization (yes vs no). Patients are randomized to 1 of 2 treatment arms.

    * Arm I: Patients receive MDX-010 in the same manner as the HLA-A*0201-negative patients.
    * Arm II: Patients receive MDX-010 as in arm I. Patients also receive gp100:209-217 and gp100:280-288 peptides emulsified in Montanide ISA-51 subcutaneously immediately after each MDX-010 infusion.
* Part II:

  * HLA-A*0201-negative patients (closed as of 3/7/2005): Patients receive MDX-010 as in part I. Treatment repeats every 3 weeks for up to 4 doses (2 courses of 2 escalating doses, beginning with a higher dose level than in part I) in the absence of disease progression or unacceptable toxicity.
  * HLA-A*0201-positive patients: Patients are stratified and randomized as in part I.

    * Arm I: Patients receive MDX-010 in the same manner as the HLA-A*0201-negative patients.
    * Arm II: Patients receive MDX-010 as in arm I. Patients also receive gp100:209-217 and gp100:280-288 peptides emulsified in Montanide ISA-51 subcutaneously immediately after each MDX-010 infusion.

In both parts, patients with stable disease or a complete response (CR) after completing all courses of MDX-010 may receive 1 additional course of therapy in the absence of unacceptable toxicity. Patients achieving a partial response may continue to recieve treatment with MDX-010 at the same dose, in the absence of unacceptable toxicity, until CR or until tumor is no longer shrinking.

Patients are followed at 3 weeks, every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 35-179 patients (up to 35 for part I [closed as of 3/7/05] and 69-141 [23-47 per arm (arm I closed as of 3/7/05)] for part II) will be accrued for this study within 3-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV melanoma
* Clinically evaluable or measurable disease
* No mucosal or ocular melanoma

PATIENT CHARACTERISTICS:

Age

* 16 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 6 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Hematocrit ≥ 28%
* WBC ≥ 2,500/mm^3

Hepatic

* AST ≤ 3 times upper limit of normal (ULN)
* Bilirubin ≤ ULN (< 3 mg/dL for patients with Gilbert's syndrome)
* Hepatitis B surface antigen negative
* Hepatitis C virus antibody negative

Renal

* Creatinine < 2 mg/dL

Immunologic

* HIV negative
* No history of any of the following:

  * Inflammatory bowel disease
  * Regional enteritis
  * Connective tissue disorders (e.g., systemic lupus erythematosus)
  * Rheumatoid arthritis
  * Autoimmune inflammatory eye disease
  * Sjögren's syndrome
  * Inflammatory neurologic disorder (e.g., multiple sclerosis)
* No active infection
* No active autoimmune disease that may cause life-threatening symptoms or severe organ/tissue damage

  * Vitiligo, autoimmune thyroiditis, or skin rashes associated with prior therapy are allowed if patient has recovered to grade 1 or less toxicity
* No systemic hypersensitivity to study agents

  * Prior local reaction (e.g., delayed hypersensitivity or glaucomatous reactions) to Montanide ISA-51 or gp100 injections allowed
* No autoimmune disease requiring active therapy with any form of steroid or immunosuppressant

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No concurrent underlying medical condition that would preclude study participation
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody
* Prior therapy with gp100 peptides or any other immunotherapy allowed

Chemotherapy

* At least 6 weeks since prior nitrosoureas and recovered (toxicity no greater than grade 1)
* No concurrent chemotherapy

Endocrine therapy

* At least 4 weeks since prior steroids
* No concurrent systemic, inhaled, optical, or topical corticosteroids

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 3 weeks since prior systemic therapy for melanoma and recovered (toxicity no greater than grade 1)
* No concurrent immunosuppressive agents (e.g., cyclosporine)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 179 (Estimated)
Dates: Start 2004-03; Primary Completion 2007-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Objective response (partial and complete)

SECONDARY OUTCOMES:
Safety
Immune response activity

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Principal Investigator — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Schadendorf D, Hodi FS, Robert C, Weber JS, Margolin K, Hamid O, Patt D, Chen TT, Berman DM, Wolchok JD. Pooled Analysis of Long-Term Survival Data From Phase II and Phase III Trials of Ipilimumab in Unresectable or Metastatic Melanoma. J Clin Oncol. 2015 Jun 10;33(17):1889-94. doi: 10.1200/JCO.2014.56.2736. Epub 2015 Feb 9. PMID 25667295